CLINICAL TRIAL: NCT01161836
Title: An Open-label Study Investigating the Disposition and QT/QTc Interval Effects of 400 mg [14C]-Iniparib(3.7 MBq, 100 µCi) Administered at Cycle 1 as a 60-minute Intravenous Infusion to Patients With Advanced Solid Tumors Followed by Extended Treatment With BSI-201 With or Without Additional Chemotherapy
Brief Title: An Open-label Study Investigating the Disposition and QT/QTc Interval Effects of 400 mg [14C]-Iniparib(3.7 MBq, 100 µCi)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEX11505; 20100109 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iniparib (Experimental): Segment 1: 400 mg [14C]-iniparib single administration
  Segment 2: Iniparib, 5.6mg/kg, extension treatment with or without additional chemotherapy
  Interventions: Drug: Iniparib

INTERVENTIONS:
Drug: Iniparib — Solution for infusion
  60-minute intravenous infusion
  Other Names: SAR240550; BSI-201

SUMMARY:
This is a Phase 1, multi-center, open-label study.

During Segment 1, patients are administered a single IV administration of [14C]-iniparib.

During Segment 2, patients are administered iniparib with or without additional chemotherapy. Acceptable chemotherapy regimens is limited to those for which previous experience with iniparib exists.

ELIGIBILITY:
Male or female patients with advanced solid tumors that are refractory to standard treatment or for which no standard treatment exists; patients must be at least 18 years old.

Additional criteria are also required and should be evaluated by the research staff.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The excretion balance and systemic exposure of radioactivity after intravenous (IV) administration of [14C]-iniparib | Up to 35 days
The pharmacokinetics of iniparib, iodo-amino-benzamide (IABM) and iodo-amino-benzoic acid (IABA) and their contribution to overall exposure of radioactivity | up to 35 days
The effects of iniparib on changes in the ECG with special focus on the QTcF interval duration | 96 hours
The metabolic pathways of iniparib and identify the chemical structures of the main metabolites. | Up to 35 days

SECONDARY OUTCOMES:
The clinical and biological tolerability of iniparib. | During treatment and until 30 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Northwest Medical Specialties, Tacoma, Washington, United States